CLINICAL TRIAL: NCT00703157
Title: Surgical or Catheter Ablations in Patients With Lone Atrial Fibrillation: Determination of Acute and Long Term Success Rate (SCALAF Success Trial)
Brief Title: Surgical or Catheter Ablation of Lone Atrial Fibrillation (AF) Patients
Acronym: SCALAF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollments slowed down significantly, despite several attempts to re-launch.
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRC-CS
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Arm 1: Catheter Ablation
  Interventions: Procedure: Catheter Ablation
- 2 (Active Comparator): Arm 2: Surgical Ablation.
  Interventions: Procedure: Surgical Ablation

INTERVENTIONS:
Procedure: Catheter Ablation — Patients undergoing left atrial circumferential pulmonary vein ostia ablation.
  Arms: 1
Procedure: Surgical Ablation — patients undergoing left atrial circumferential pulmonary vein ostia ablation via minimal invasive surgery.
  Arms: 2

SUMMARY:
Prospective randomized interventional trial comparing the efficacy of circumferential pulmonary vein ostia ablation using surgical versus catheter techniques in the treatment of paroxysmal atrial fibrillation. Success rate determined by REVEAL-XT (AF implantable monitoring device).

DETAILED DESCRIPTION:
Title: Surgical or Catheter Ablation in patients with Lone Atrial Fibrillation: determination of acute and long term SUCCESS (SCALAF-success trial).

Background: Anti-arrhythmic drugs are used in daily practice to treat patients with paroxysmal idiopatic AF. Often the origin of the AF can be found in the muscle sleeves running up the pulmonary veins. Drug treatment is not always successful and prone to evoke negative side effects. The surgical MAZE procedure was applied in the past, but this is a time consuming, cumbersome technique, often associated with significant complications. Cardiac radio-frequency ablation offers an alternative, easy and less time consuming treatment: lesions prevent normal electrical wave front propagation and might stop the continuation of atrial fibrillation wave fronts. Ablation can be implemented by use of special catheters inserted via the groin or using the Medtronic Cardioblate® Surgical Ablation System applied via minimal invasive surgical techniques.

Purpose: Compare the effectiveness of pulmonary vein isolation achieved via catheter or via surgical ablation techniques to treat patients with paroxysmal lone AF.

Study design: A prospective, randomized multi-center interventional study.

Patients: Patients suffering from paroxysmal idiopatic AF (no associated or underlying structural heart disease) complying with following inclusion criteria:

* minimally one documented AF-episode in the last 6 months;
* refractory to at least 2 class I or III anti-arrhythmic drugs;
* age > 18 year

Intervention: Patients are randomized to either the surgical or the catheter ablation group and receive the indicated treatment. During the critical assessment period, the patients are weaned from anti-arrhythmic medication.

Primary endpoint: Reduction in AF occurrence measured by the AF-burden parameter in the critical period between 3 and 6 months post-ablation. AF burden is measured automatically by means of the Reveal XT, implanted at study enrolment to document the baseline characteristics.

Secondary endpoints:

* Failure of therapy requiring re-interventions;
* Duration, burden and costs of ablation procedures:
* Reduction in frequency, duration and level of severity of AF symptoms;
* Occurences of treatments of arrythmic episodes;
* Assessment of AF burden during follow-up period
* Symptoms associated with AF;
* Reduced necessity of anti-arrhythmic or anticoagulant medication;
* Left atrial dimensions and contractility
* Adverse events associated with the ablation therapy;
* Occurrence of other clinical adverse events (TIA, CVA, bleeds, tamponade, MI) at 3, 6, 12 and 24 months of follow up
* Mortality and hospitalisation

Risk assessment: Possible side effects : irregular heart rhythm, pericardial fluid, stroke, heart infarct, disturbances of the conduction system in the heart, local pain at the site of incisions, heart failure or reduced pump function of the heart.

Possible benefits: Regulation of the heart rhythm without applying MAZE procedure or opening of the thorax. Reduction or relief from symptoms associated with AF. Partial or complete reduction of anti-arrhythmic medication. Control of anti-coagulant medication. Improved quality of life for the patients.

Visits are planned at study entrance and Reveal XT implant (assessment at baseline, application of the ablation therapy), discharge from hospital, and at 3, 6, 12 and 24 months post-ablation.

ELIGIBILITY:
Inclusion Criteria:

* Patient has documented Paroxysmal AF as defined by the ACC/AHA/ESC guidelines
* Minimal one documented AF episode in the last 6 months
* Refractory to minimal two Class I or III anti-arrhythmic drug
* Age > 18 years
* Signed and dated the Patient Informed Consent.
* Patient can tolerate anti-coagulation therapy (Warfarin/Coumadin)

Exclusion Criteria:

* Patient has a structural heart disease
* Ejection fraction < 40 %
* Echocardiographic evidence for a left atrium > 45 mm (parasternal axis)
* Patients on amiodarone, or patients known to be intolerant for amiodarone
* Dextrocardia, current endocarditis, systemic infection, renal failure
* Patient has known cerebrovascular disease, including a history of stroke, CVA or TIA
* Pregnancy at enrolment; or planned pregnancy within the follow up period
* Patient has a life expectancy less than 1 year
* The subject is participating in another device or drug study
* The patient is unable and/or unwilling to cooperate with study procedures or required follow up visits
* Echocardiographic (TTE) evidence for presence of left atrial thrombus
* Previous (cardio-) thoracic surgery
* Previous left atrial ablation
* Patients with permanent or persistent AF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-11; Primary Completion 2015-08 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hauw Sie, MD, Principal Investigator — Isala
Locations (1):
- Isala Klinieken, Zwolle, Netherlands

IPD SHARING:
Plan to Share IPD: No
There is no plan or intention to share individual participant data (IPD)

REFERENCES:
- [Derived] Buist TJ, Adiyaman A, Beukema RJ, Smit JJJ, Delnoy PPHM, Hemels MEW, Sie HT, Ramdat Misier AR, Elvan A. Quality of life after catheter and minimally invasive surgical ablation of paroxysmal and early persistent atrial fibrillation: results from the SCALAF trial. Clin Res Cardiol. 2020 Feb;109(2):215-224. doi: 10.1007/s00392-019-01504-z. Epub 2019 Jun 24. PMID 31236689
- [Derived] Adiyaman A, Buist TJ, Beukema RJ, Smit JJJ, Delnoy PPHM, Hemels MEW, Sie HT, Ramdat Misier AR, Elvan A. Randomized Controlled Trial of Surgical Versus Catheter Ablation for Paroxysmal and Early Persistent Atrial Fibrillation. Circ Arrhythm Electrophysiol. 2018 Oct;11(10):e006182. doi: 10.1161/CIRCEP.118.006182. PMID 30354411

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eighty (80) subjects were enrolled, of whom 52 were randomized. A Reveal XT Implantable device was implanted in all subjects after Informed Consent. The subjects were followed for a minimum of 1 week and a maximum of 6 months. If the subject demonstrated a minimum of 10% AF burden during this period and had complaints, the subject was randomized.
Groups:
- Catheter: Catheter Ablation
- Surgery: Surgical Ablation
Period: Overall Study
Arm/Group | Catheter | Surgery
Started | 26 | 26
6 Months FU | 25 | 25
24 Months FU | 22 | 24
Completed | 22 | 24
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — source data permanently lost/ other | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Catheter | Surgery | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (7) | 55 (9) | 58 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 20 | 21 | 41
NYHA Class [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Functional Classification places patients in one of four categories based on their limitations during physical activity.The limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina.
  Class I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  Class II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  Participants
    I | 25 | 23 | 48
    II | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in AF Burden After Ablation Therapy Measured With REVEAL-XT Implantable Device.
Description: AF Burden is defined as the percentage of time during the follow-up period that a subject is in AF, as measured by the REVEAL-XT implantable device.
Time Frame: Baseline through 3-6 months post-ablation
Measure: Mean (Standard Deviation); unit: percentage of time in AF
Groups:
- All Subjects: All Subjects, regardless of randomization group
Arm/Group | Catheter | Surgery | All Subjects
Number analyzed (Participants) | 24 | 26 | 50
percentage of time in AF
  Pre-ablation | 7.6 (7.4) | 7.9 (8.7) | 7.8 (8.0)
  Blanking Period | 1.6 (4.2) | 3.6 (6.1) | 2.6 (5.3)
  Absolute Change Pre to Blanking | -6.0 (6.1) | -4.3 (7.2) | -5.1 (6.7)
  Post-Ablation | 0.5 (1.4) | 2.0 (5.5) | 1.3 (4.1)
  Absolute Change Blanking to Post | -1.1 (3.2) | -1.1 (5.5) | -1.3 (4.5)
  Percent Change Pre to Post | -77.8 (68.4) | -70.8 (65.1) | -74.2 (66.1)
  Absolute Change Pre to Post | -7.1 (7.1) | -5.8 (9.1) | -6.5 (8.1)

2. Secondary Outcome: Treatment Failures Requiring Redo or Alternative Therapy
Time Frame: Time from procedure until 6 months post-ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Catheter | Surgery | All Subjects
Number analyzed (Participants) | 26 | 26 | 52
Participants | 5 | 0 | 5

3. Secondary Outcome: Number of Subjects With Adverse Events, Associated With the Ablation Procedure
Time Frame: Time from procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Catheter | Surgery | All Subjects
Number analyzed (Participants) | 26 | 26 | 52
Participants | 5 | 16 | 21

4. Secondary Outcome: Mortality and Hospitalization
Time Frame: Time from procedure until 24 months post-ablation
Measure: Number; unit: participants
Arm/Group | Catheter | Surgery | All Subjects
Number analyzed (Participants) | 26 | 26 | 52
participants
  Any Hospitalization | 24 | 31 | 55
  Any Procedure-Related Hospitalization | 5 | 9 | 14
  Death | 0 | 1 | 1

5. Secondary Outcome: Duration, Burden and Costs of Treatment Procedures
Time Frame: Through 24 months post- ablation
Population: Data were not collected
Arm/Group | Catheter | Surgery
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Reduced Number, Duration and Severity of AF Symptoms
Time Frame: Through 24 months post-ablation
Population: Data were not collected
Arm/Group | Catheter | Surgery
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Symptoms Associated With Atrial Arrhythmias
Time Frame: Through 24 months post-ablation
Population: Data were not collected
Arm/Group | Catheter | Surgery
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Occurences of Treatment of Arrhythmic Episodes
Time Frame: Through 24 months post-ablation
Population: Data were not collected
Arm/Group | Catheter | Surgery
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Assessment of AF Burden
Time Frame: Through 24 months post-ablation
Population: Data were not collected
Arm/Group | Catheter | Surgery
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Reduced Anti-arrhythmic Drug Requirement
Time Frame: Through 24 months post-ablation
Population: Data were not collected
Arm/Group | Catheter | Surgery
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Left Atrial Dimension and Contractility
Time Frame: Through 24 months post-ablation
Population: Data were not collected
Arm/Group | Catheter | Surgery
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse Events were monitored for a limited timeframe, ie.up to 6 Months Post-Ablation, by Randomization Group
Groups:
- All Randomized Subjects: All Randomized Subjects, regardless of randomization group
Arm/Group | Catheter | Surgery | All Randomized Subjects
All-Cause Mortality (participants affected / at risk) | 0/26 | 1/26 | 1/52
Serious Adverse Events (participants affected / at risk) | 10/26 | 15/26 | 25/52
Other Adverse Events (participants affected / at risk) | 3/26 | 8/26 | 11/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheter (N=26) | Surgery (N=26) | All Randomized Subjects (N=52)
Atrial Fibrillation (Cardiac disorders) | 5 (9) | 1 (1) | 6 (10)
Cerebralvascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Postoperative fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 2 (2)
Arteriospasm coronary (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (3) | 3 (4)
Chest Pain (General disorders) | 0 (0) | 2 (2) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
External Cephalic Version (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Parapalegia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 1 (1) | 1 (1) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Blindness transient (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Dressler's syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Sternotomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheter (N=26) | Surgery (N=26) | All Randomized Subjects (N=52)
Atrial Fibrillation (Cardiac disorders) | 3 (5) | 6 (6) | 9 (11)
Pericarditis (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
The study stopped early, prior to meeting the target number of subjects per group. The reported results and conclusions are based on these limited data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less